CLINICAL TRIAL: NCT04965766
Title: Phase 2, Open Label Study of Patritumab Deruxtecan (U3-1402), an Anti-HER3-Antibody Drug Conjugate (ADC), in Patients With Advanced Breast Cancer, With Biomarker Analyses to Characterize Response to Therapy
Brief Title: Patritumab Deruxtecan (U3-1402) in Unresectable Locally Advanced or Metastatic Breast Cancer
Acronym: ICARUS BREAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-005722-28; 2020/3188 (Other: CSET number); 2023-505923-30-00 (EU CTIS Number)
Record Dates: First submitted 2021-06-03; First posted 2021-07-16 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer
Keywords: Metastatic breast cancer; Advanced breast cancer; Unresectable breast cancer; HER2- Breast Cancer; Hormone-receptor positive breast cancer; HR+ breast cancer; Antibody drug conjugate; ADC; Patritumab deruxtecan; U3-1402; Refractory metastatic breast cancer; HER2 Negative; MBC; ABC; Metastatic BC; Advanced BC; Unresectable BC; Refractory advanced breast cancer; Refractory ABC; Refractory MBC; HER3-DXd; estrogen receptor positive; progesterone receptor positive; ER+; PR+; ER+/PR+
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Intervention Model Description: One group of 139 participants treated with U3-1402
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U3-1402 (Experimental): All participants enrolled in the study will receive U3-1402 at a dose of 5.6 mg/kg every 3 weeks until progression or until unacceptable toxicity
  Interventions: Drug: U3-1402

INTERVENTIONS:
Drug: U3-1402 — U3-1402 is uniquely designed to target HER3-a receptor that contributes to treatment resistance and poor prognosis in hormone receptor-positive, HER2-negative (HR+/HER2-) breast cancer patients. This drug is distinct from other interventions due to its composition as an antibody-drug conjugate (ADC): a monoclonal antibody against HER3 conjugated to a topoisomerase I inhibitor, which specifically targets HER3-overexpressing tumor cells. The drug is delivered via a cleavable linker that allows for controlled release of the chemotherapeutic agent within the cancer cells, minimizing systemic side effects.
  Other Names: HER3-DXd

SUMMARY:
This study aims to evaluate the efficacy and safety of U3-1402 in participants with advanced breast cancer (ABC). Participants have to be hormone-receptor positive (HR+) and have to be resistant to endocrine therapy and cyclin-dependent kinases 4 and 6 (CDK4/6) inhibitors. Participants may have received multiple lines of endocrine therapy with or without targeted therapies and must have received only one line of chemotherapy for ABC.

Moreover, the immune effects, the predictors of resistance and response to treatment, the effect of the chemotherapy on deoxyribonucleic acid (DNA) replication will be assessed and will help identify the subgroups that will mostly benefit from the treatment. The pharmacokinetics of the product and the anti-drug antibody (ADA) will be also evaluated.

A total of 99 participants are planned to be treated in the study. Participants will receive, every three weeks, a dose of U3-1402 equivalent to 5.6 mg/kg of body weight until progression or until unacceptable toxicity.

Tumor evaluation will be performed every six weeks by the mean of a computed tomography for the thorax, abdomen and pelvis (TAP CT-scan) or a magnetic resonance imaging (MRI). Brain and/or bone CT scans will be also performed throughout the study for participants with brain and/or bone metastasis. A PET scan combined with contrast enhanced CT scan can replace all the above-mentioned imaging if performed at baseline considering that the same imaging technique should be used throughout the study.

The safety of the product will be assessed at each cycle, through complete clinical exams, biological tests, electrocardiograms (ECGs), cardiac echographies (ECHOs) and through the collection of ongoing toxicities or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults with histologically-confirmed HER2 negative, unresectable locally advanced or metastatic breast cancer that is hormone receptor positive (HR+) at the time of the first breast cancer diagnosis
* Participants with a documented radiologic unresectable or metastatic progression
* Participants may have received anthracyclines and taxanes as (neo) adjuvant treatment and must have received one line of chemotherapy for Advanced breast cancer (ABC), but not more than one line. Participants must have a clinically or radiologically documented evidence of tumor progression on or after cyclin dependent kinase 4/6 (CDK 4/ 6) inhibitor combined with endocrine therapy. Previous treatments with PI3K inhibitors, mTOR inhibitors, AKT-inhibitors and poly ADP ribose polymerase (PARP)-inhibitors are allowed
* Participants must have a tumor site easily accessible to biopsy (with exception of bone metastasis)
* Participants must have at least one radiologically measurable lesion (different from the biopsy site)
* Participants must have an ECOG PS equals to 0 or 1
* Participants must have a life expectancy of 12 weeks or more
* Participants must have adequate bone marrow reserve and organ function, based on local laboratory data within 14 days prior to Cycle 1, Day 1
* Female patients of reproductive/childbearing potential must have a negative pregnancy test at screening (serum test within 14 days or urine test within 72 hours of enrollment). A positive urine pregnancy test result must be confirmed by a serum test. Patients must agree to use a highly effective form of contraception or avoid intercourse during and upon completion of the study and for at least 7 months after the last dose of study drug.

The following contraception methods are considered highly effective:

1. Hormonal or nonhormonal intrauterine device (IUD)
2. Progestogen-only subdermal contraceptive implant
3. Bilateral tubal occlusion
4. Vasectomized partner
5. Complete sexual abstinence defined as refraining from heterosexual intercourse during and upon completion of the study and for at least 7 months for females after the last dose of study drug.

Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception. Penile/external condoms for male partners must be used in addition to the female patient's hormonal contraception for the duration treatment intervention and until 7 months following the last dose of trial intervention. Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 7 months after the final study drug administration.

* A male participant capable of producing sperm is eligible to participate if he agrees to the following during the intervention period and for at least the time needed to eliminate each trial intervention. The length of time required to continue contraception after last dose for each trial intervention is 4 months. Avoid donating sperm. Note: Preservation of sperm should be considered prior to enrollment/randomization in this trial. Use a penile/external condom when having penile-vaginal intercourse with a nonparticipant of childbearing potential, PLUS partner use of an additional contraceptive method (see below), as a condom may break or leak:

  1. Progestogen-only contraceptive implant
  2. Hormonal or nonhormonal IUD
  3. Bilateral tubal occlusion (includes tubal ligation)
  4. Combined (estrogen- and progestogen-containing) hormonal contraception (oral, intravaginal, transdermal, injectable)
  5. Progestogen-only hormonal contraception (oral, injectable)
  6. Progesterone-only hormonal contraception where inhibition of ovulation is not the primary mode of action
  7. Cervical cap, diaphragm, or sponge with spermicide Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

     If the contraception requirements in the local label for any of the trial interventions are more stringent than the requirements above, the local label requirements are to be followed. Note: If the participant is azoospermic (vasectomized or secondary to medical cause, documented from the site personnel's review of the participant's medical records, medical examination, or medical history interview), no contraception is required.

     Male participants must not freeze or donate sperm starting at screening and throughout the study period, and for at least 4 months after the final study drug administration
* Participant must understand, sign, and date the written ICF prior to any protocol-specific procedures performed. Participant should be able and willing to comply with study visits and procedure as per protocol
* Participant must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Breast cancer amenable for resection or radiation therapy with curative intent
* Any history of interstitial lung disease (ILD), actual ILD, or a suspicion of an ILD
* Clinically severe pulmonary compromise (based on investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

  1. Any underlying pulmonary disorder
  2. Any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement
  3. OR prior pneumonectomy
* The use of chronic systemic corticosteroids at a dose superior to 10 mg daily of prednisone or equivalent or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Participants who require use of bronchodilators, inhaled steroids, or local steroid injections may be included in the study
* Evidence of any leptomeningeal disease
* Evidence of corneal disease
* Any evidence of severe or uncontrolled systemic diseases including active bleeding diatheses, active infection, psychiatric illness/social situations, geographical factors, substance abuse, or other factors which in the investigator's opinion makes it undesirable for the participant to participate in the study or which would jeopardize compliance with the protocol
* Evidence of clinically active spinal cord compression or brain metastases defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms
* Exposure to prior systemic anticancer therapy (including investigational agents) within 4 weeks or 5 half-lives (whichever is shorter) before enrollment.
* Inadequate washout period prior to Cycle 1 Day 1, defined as:

  1. Whole brain radiation therapy <14 days or stereotactic brain radiation therapy <7 days.
  2. Immune checkpoint inhibitor therapy <21 days
  3. Hormonal therapy <21 days
  4. Major surgery (excluding placement of vascular access) <28 days.
  5. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days.
  6. Chloroquine or hydroxychloroquine ≤ 14 days
  7. Live virus vaccination <28 days.
* Prior treatment with an anti-HER3 antibody and/or ADC containing an exatecan derivative that is a topoisomerase I inhibitor
* Participants with a grade equals or greater than 2 unresolved toxicities from previous anticancer therapy (other than alopecia)
* A history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of U3-1402, or to other monoclonal antibodies
* Any evidence of primary malignancy other than locally advanced or metastatic lung cancer within three years prior to Cycle 1 Day 1, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated
* Uncontrolled or significant cardiovascular disease prior to Cycle 1 Day :

  1. Corrected QT interval higher than 470 ms for females and 450 ms for males according to Fridericia's formula (QTcF) and assessed based on triplicate ECGs, approximately 1 minute apart
  2. Left ventricular ejection fraction (LVEF) less than 50% by either ECHO or cardiac MRI or multigated acquisition scan (MUGA)
  3. Resting systolic blood pressure higher than 140 mmHg or diastolic blood pressure higher than 90 mmHg
  4. Myocardial infarction within six months
  5. Symptomatic congestive heart failure (NYHA Classes 2 to 4 within 28 days before treatment)
  6. Uncontrolled angina pectoris within six months.
  7. Cardiac arrhythmia requiring antiarrhythmic treatment
* Evidence of active or uncontrolled hepatitis B virus infection (HBV)

Participants are eligible:

1. If HBsAg positive with chronic HBV infection (lasting 6 months or longer) and meet conditions below:

   * HBV DNA viral load <2000 IU/mL
   * Start or maintain antiviral treatment if clinically indicated as per the investigator.
2. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT <3 × ULN, which are not attributable to HBV infection - Evidence of active or uncontrolled hepatitis C virus infection (HCV).

Participants are eligible if:

1. History of hepatitis C infection eligible if the HCV viral load is below the level of detection in the absence of antiviral therapy during the previous 4 weeks
2. Have normal transaminase values, or, if liver metastases are present, abnormal transaminases with a result of AST/ALT < 3 × ULN, which are not attributable to HCV infection - Evidence of active or uncontrolled human immunodeficiency virus (HIV infection. Subjects must be tested for HIV viral load during the Screening Period if acceptable by local regulations or IRBs/IECs.

Participants are eligible if:

1. CD4+ T-cell count ≥350 cells/mm3 at the time of screening 16
2. Virologic suppression defined as confirmed HIV RNA level below 50 or the LLOQ (below the limit of detection) at the time of screening and for at least 12 weeks before screening
3. No AIDS-defining opportunistic infections or conditions within the past 12 months
4. On stable ART regimen, without changes in drugs or dose modification, for at least 4 weeks before trial entry (Day 1) and agree to continue ART throughout the trial.

   * Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's judgment, could affect the safety of the subject; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results.
   * Evidence of ongoing uncontrolled systemic bacterial, fungal, or viral infection. Subjects with localized fungal infections of skin or nails are eligible.
   * Female patient who is pregnant or breastfeeding or intends to become pregnant during the study.
   * Patient with any psychological, familial, sociological or geographical condition potentially hindering compliance with the study protocol procedures and follow-up schedule.
   * Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
   * Participation in another clinical trial evaluating an experimental drug (except non-interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2030-04-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of objective response rate (ORR) based on investigator assessment | During treatment period, an average of 8 months
  Defined as the proportion of participants who achieved a confirmed complete response (CR) or partial response (PR) assessed by investigators

SECONDARY OUTCOMES:
Evaluation of duration of response (DOR, investigator-assessed and as per retrospective central review) | From cycle 3 (Week 6) up to 3 years after the EoT, an average of 42 months
  Applicable to participants with either complete response (CR) or partial response (PR) and is defined as the time from the first documented CR or PR until the date of disease progression, or until the date of death. It will be evaluated in the overall population and in subgroups of patients according to investigator assessment and as per retrospective central review
Evaluation of progression free Survival (PFS), investigator-assessed and as per retrospective central review | From cycle 3 (Week 6) up to 3 years after the EoT, an average of 42 months
  Defined as the time date of the first dose until progression or death from any cause, whichever occurs first. It will be evaluated in the overall population according to investigator assessment and as per retrospective central review
Evaluation of clinical benefit ratio (CBR), investigator-assessed and as per retrospective central review | From cycle 3 (Week 6) up to 3 years after the EoT, an average of 42 months
  Defined as the presence of at least a PR or CR, or a stable disease (SD) for more than six months under treatment. It will be evaluated in the overall population according to investigator assessment and as per retrospective central review
Percentage of patients experiencing adverse events | During treatment (at each cycle), at EoT and up to 47 days after EoT, an average of 9 months
Frequency of treatment emergent adverse events (TEAEs) leading to change in treatment dose | During treatment, an average of 8 months
Incidence of abnormal laboratory test results | During treatment (at each cycle) and at EoT an average of 8 months
Incidence of abnormal ECG readings | During treatment and at EoT an average of 8 months
Physical functioning sub-scale score of the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) based on a scale from 1 to 4, where higher scores mean worse outcome | During treatment (Cycles 1, 2, 3 and then every 2 cycles), at EoT and then up to 3 years after EoT, an average of 42 months
Changes in Eastern Cooperative Oncology Group performance status [ECOG PS] based on a score from 1 to 5, where higher scores mean worse outcomes | During treatment (at each cycle) and at EoT, an average of 8 months
Change in left ventricular ejection fraction (LVEF) | During treatment and at EoT, an average of 8 months
Global health sub-scale score of the European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) based on a scale from 1 to 7, where higher scores mean better outcome | During treatment (Cycles 1, 2, 3 and then every 2 cycles), at EoT and up to 3 years after EoT, an average of 42 months
Severity of adverse events as assessed by CTCAE v5. | During treatment (at each cycle), at EoT and up to 47 days after EoT, an average of 9 months
Objective response rate (ORR) as per central retrospective review | During treatment period, an average of 8 months
  Defined as the proportion of participants who achieved a confirmed complete response (CR) or partial response (PR) assessed by investigators and as per central retrospective review
Overall survival (OS) | From C1D1 until death, an average of 42 months
  Defined as the time from date of first dose until death. Patients alive at last follow-up will be censored at this date.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara PISTILLI, Dr, Study Director — Gustave Roussy, Cancer Campus, Grand Paris
Locations (11):
- France (11):
  - Centre Georges François Leclerc, Dijon
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hôpital Tenon, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Pistilli B, Mosele F, Corcos N, Pierotti L, Pradat Y, Le Bescond L, Lacroix-Triki M, Nachabeh G, Alfaro A, Catelain C, Job B, Mami-Chouaib F, Badel S, Farace F, Oulhen M, Kannouche P, Tran DTN, Droin N, Vicier C, Frenel JS, D'Hondt V, Dalenc F, Bachelot T, Ducoulombier A, Benderra MA, Loirat D, Mayeur D, Deluche E, Deneuve J, Cheikh-Hussin R, Guyader P, Signolle N, Godefroy K, Talbot H, Vakalopoulou M, Christodoulidis S, Bernard E, Koudou Y, Sporchia A, Suto F, Li L, Sternberg DW, Michiels S, Andre F, Sellami D, Montagnac G. Patritumab deruxtecan in HR+HER2- advanced breast cancer: a phase 2 trial. Nat Med. 2025 Oct;31(10):3492-3503. doi: 10.1038/s41591-025-03885-3. Epub 2025 Sep 4. PMID 40908353